CLINICAL TRIAL: NCT06756009
Title: Evaluation of Chronic Liver Disease Condition and Transplant Prognosis Assisted by Eye Biological Parameters
Status: Recruiting | Type: Observational
Sponsor: Zhongshan Ophthalmic Center, Sun Yat-sen University (Other)
Collaborators: First Affiliated Hospital, Sun Yat-Sen University (Other); Second Affiliated Hospital, Sun Yat-Sen University (Other); Guangdong Provincial People's Hospital (Other); Nanfang Hospital of Southern Medical University, Guangdong of China (Unknown); Zhongshan People's Hospital, Guangdong, China (Other); Guangdong Provincial People's Hospital, China (Unknown); First People's Hospital of Foshan (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Zhongshan Ophthalmic Center, Sun Yat-sen University
Other Study IDs: 2021KYPJ148
Record Dates: First submitted 2024-12-25; First posted 2025-01-01 (Actual); Last update posted 2025-01-01 (Actual); Status verified 2024-08

CONDITIONS: Diagnostic Techniques, Ophthalmological; Liver Transplantation; Liver Cirrhoses
Keywords: Diagnostic Techniques, Ophthalmological; liver transplantation; Liver Cirrhoses

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- preoperative group: Registered liver transplant patients from preoperative to postoperative follow-up
  Interventions: Diagnostic Test: Ophthalmic examination; Diagnostic Test: General Condition Examination
- Simple postoperative group: Follow up from after liver transplantation
  Interventions: Diagnostic Test: Ophthalmic examination; Diagnostic Test: General Condition Examination
- Healthy control group: Healthy individuals without liver disease
  Interventions: Diagnostic Test: Ophthalmic examination; Diagnostic Test: General Condition Examination

INTERVENTIONS:
Diagnostic Test: Ophthalmic examination — Various ophthalmic examination modalities, including slit lamp photography, fundus photography, optical coherence tomography imaging and optical coherence tomography angiography, etc.
Diagnostic Test: General Condition Examination — Various general condition examination, including blood pressure measurement, blood glucose testing, blood routine examination, coagulation function test, liver function test, etc.

SUMMARY:
This study investigates the correlation between ocular biological characteristics and overall conditions before and after liver transplantation by collecting ocular biological characteristics. Explore whether it is possible to construct a clinical prediction model for liver transplantation by incorporating ocular biometric features, in order to optimize disease management before and after liver transplantation.

DETAILED DESCRIPTION:
This study is a bidirectional cohort study, which retrospectively analysed data from a prospective database to construct a model, and prospectively collected patient information from preoperative to postoperative for model improvement and validation.

ELIGIBILITY:
Inclusion Criteria:

1. Age greater than or equal to 18 years old;
2. Late stage liver disease patients waiting for liver transplantation treatment, as well as patients with varying degrees of cirrhosis;
3. Can collect complete basic demographic information, liver function blood test indicators, liver pathology and imaging examination results;
4. Can cooperate with eye OCT, OCTA and other examinations, and obtain qualified examination parameters;
5. Voluntarily follow the clinical trial protocol and sign the informed consent form.

Exclusion Criteria:

1. History of other organ transplant surgeries;
2. History of intraocular laser treatment, medication injection, and surgery;
3. History of high myopia, glaucoma, and retinal choroidal related eye diseases;
4. History of major systemic diseases other than liver disease;
5. Individuals whose overall body and eye conditions cannot cooperate with eye examinations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The liver transplant population was recruited from individuals who went to cooperative medical unit for liver transplant registration, while normal individuals were recruited from the project responsible unit.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The performance of predicting the prognosis of liver transplantation | 1 week and 1 year after liver transplantation
  Based on the outcomes of early graft dysfunction and 1-year graft survival rate, the area under the receiver operating characteristic curve, specificity, and sensitivity of the model

SECONDARY OUTCOMES:
The performance of the model in assessing the severity of liver disease | 1 year
  The confusion matrix of the model based on the MELD score results

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No